CLINICAL TRIAL: NCT06966024
Title: An Open-label, Phase 1 Study of DCC-2812 Monotherapy in Participants With Advanced or Metastatic Renal Cell Carcinoma, Urothelial Cancer, or Castration-Resistant Prostate Cancer
Brief Title: Study of DCC-2812 in Participants With Advanced Genitourinary Cancers
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Deciphera Pharmaceuticals, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DCC-2812-01-001
Record Dates: First submitted 2025-05-02; First posted 2025-05-11 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Renal Cell Carcinoma; Urothelial Carcinoma; Castration-resistant Prostate Cancer
Keywords: Advanced malignancies
MeSH Terms: conditions — Carcinoma, Renal Cell; Carcinoma, Transitional Cell

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- DCC-2812 (Experimental): Participants will receive DCC-2812 in dose escalation manner per dosing regimen depending upon evolving pharmacokinetic (PK), pharmacodynamic, and safety data.
  Interventions: Drug: DCC-2812

INTERVENTIONS:
Drug: DCC-2812 — Administered orally

SUMMARY:
This is a multicenter clinical trial to evaluate the safety and preliminary activity of the selective general control nonderepressible 2 (GCN2) activator DCC-2812 as monotherapy in advanced/metastatic renal cell carcinoma (RCC), urothelial carcinoma, and castration-resistant prostate cancer.

ELIGIBILITY:
Key Inclusion Criteria:

* Have confirmed Advanced or Metastatic Renal Cell Carcinoma, Urothelial Cancer, or Castration-Resistant Prostate Cancer
* Able to take oral medication
* If a female is of childbearing potential, must have a negative pregnancy test prior to enrollment and all participants agree to follow the contraception requirements
* Adequate organ function and electrolytes

Key Exclusion Criteria:

* Received any prior anticancer therapy or any investigational therapy within a specified timeframe prior to first dose of DCC-2812
* Impaired cardiac function
* Major surgery within 28 days of the first dose of study drug

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-08-27 (Actual); Primary Completion 2029-02 (Estimated); Study Completion 2029-02 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Dose-limiting Toxicities (DLTs) | Cycle 1 (28 days)
Number of Participants With Treatment-emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) | Up to 42 months
Number of Participants With Dose Reduction, Interruption, or Discontinuation of Study Drug Due to TEAEs | Up to 42 months

SECONDARY OUTCOMES:
Radiographic Objective Response Rate (rORR) per Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 42 months
Radiographic Duration of Response (rDOR) per RECIST v1.1 | Up to 42 months
PK: Maximum Observed Plasma Drug Concentration (Cmax) | Predose up to 24 hours postdose (up to 42 months)
PK: Time to Reach Cmax (Tmax) | Predose up to 24 hours postdose (up to 42 months)
PK: Area Under the Plasma Concentration-time Curve (AUC) | Predose up to 24 hours postdose (up to 42 months)
PK: Trough Plasma Concentration (Ctrough) | Predose up to 24 hours postdose (up to 42 months)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Team, Study Director — Deciphera Pharmaceuticals, LLC
Locations (3):
- United States (3):
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - NEXT Oncology, Austin, Austin, Texas
  - NEXT Oncology, San Antonio, San Antonio, Texas